CLINICAL TRIAL: NCT03262844
Title: Efficacy and Safety of Nerve Root Axial Decompression Surgery in The Treatment of Tethered Cord Syndrome: A Conservative Treatment- Controlled, Randomized, Clinical Study
Brief Title: Efficacy and Safety of Nerve Root Axial Decompression Surgery in The Treatment of Tethered Cord Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Jiangang Shi, Chief of No.2 department of spinal surgery, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CZ1702TCS
Record Dates: First submitted 2017-08-06; First posted 2017-08-25 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Tethered Cord Syndrome
MeSH Terms: conditions — Neural Tube Defects | interventions — Conservative Treatment; Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistical analysist do not know the group assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative treatment (Placebo Comparator): Conservative physiotherapy, intermittent catheterization, or drug treatment for bladder or bowel dysfunction
  Interventions: Behavioral: Conservative treatment
- Capsule surgery (Experimental): Nerve root axial decompression surgery (Capsule surgery)
  Interventions: Procedure: Capsule surgery

INTERVENTIONS:
Behavioral: Conservative treatment — The conservative treatment group will be given diet and nursing guidance, then the drug treatment or physiotherapy will be given according to the conditions of patients. Patients with bladder dysfunction will be guided to perform routine intermittent catheterization with help of their parents.
  Arms: Conservative treatment
Procedure: Capsule surgery — In the multiple segments of the spine, articular facet joint and intervertebral disc will be resected to achieve the effect of decompression.
  Specific surgical segments, osteotomy range, decompression degree of each patient needs to be designed individually.
  Arms: Capsule surgery

SUMMARY:
Background: Tethered cord syndrome (TCS) is a progressive clinical condition including a series of neurological dysfunctions and deformities attributable to abnormally increased tension on the spinal cord, which is lacking effective treatment to relieve the symptoms and prevent progression. Dr. Shi recently proposed a new technique as nerve root axial decompression surgery, which is also called capsule surgery, to treat patients with TCS. Yet, the effectiveness and safety should be further studied.

Purpose: The aim of this study is to compare the effectiveness and safety of clinical outcomes between capsule surgery and conservative treatment in patients with TCS. A study hypothesis is that outcomes will be improved after capsule surgery.

Methods: This study is a randomized clinical trial with a two-factor (2x7) research design. The TCS patients will be randomly assigned in one of the two treatment groups: capsule surgery and conservative treatment. Seven outcome measures will be collected pre-operative for baseline, and then at1, 12, 24, 48, and 96 weeks post-operative follow-up visits, including: International Consultation on Incontinence Modular Questionnaire Short Version (ICI-Q-SF), Rintala Score, a new developed Chinese version of questionnaire, Oswestry disability index (ODI), SF-12, foot function index (FFI) and Pirani score. Urodynamic testing, bladder ultrasonography, electromyogram, muscle strength and sensation of lower limbs will be obtained before and post treatment, to determine the patient's function of lower limbs. The investigator performing the outcome measures will be blinded to group assignment, and therefore will not participate in treatment. After randomization, the conservative group will be followed up in the outpatient clinic. The capsule surgery group will receive the nerve root axial decompression surgery (capsule surgery).

Data Analysis: Two 2x7 MANOVAs with repeated measures will be used to examine the differences in the seven measures between groups and at the five different time frames with the α level set at 0.05. Non-parametric tests (Mann-Whitney U tests) will be used to compare the differences in the urodynamics and muscle strength data over time and between groups.

DETAILED DESCRIPTION:
Background: Tethered cord syndrome (TCS) is a progressive clinical condition including a series of neurological dysfunctions and deformities attributable to abnormally increased tension on the spinal cord. The standard surgical treatment is untethering the spinal cord and correction of the related deformity. Although reported results are encouraging, it continues to pose challenges on management of TCS patients. Symptomatic re-tethering seems to be an inevitable result, which occurs in 20%-50% patients after untethering. Recently, filum dissection was found no good to improve urinary symptoms compared to conservative treatment in teenagers as reported in an RCT study. Also, it remained controversy when to perform the surgery and how to evaluate the benefits of surgery or conservative treatment. Dr. Shi recently proposed a new technique as nerve root axial decompression surgery, which is also called capsule surgery, to treat patients with TCS. Yet, the effectiveness and safety should be further studied.

Purpose: The aim of this study is to compare the effectiveness and safety of clinical outcomes between capsule surgery and conservative treatment in patients with TCS. A study hypothesis is that outcomes will be improved after capsule surgery.

Methods: This study is a randomized clinical trial with a two-factor (2x7) research design. The TCS patients will be randomly assigned in one of the two treatment groups: capsule surgery and conservative treatment. Seven outcome measures will be collected pre-operative for baseline, and then at1, 12, 24, 48, and 96 weeks post-operative follow-up visits, including: (1) International Consultation on Incontinence Modular Questionnaire Short Version (ICI-Q-SF) to assess the urinary functions, (2) Rintala Score for bowel function, (3) a new developed Chinese version of questionnaire to assess the quality of life in patients and parents due to bladder dysfunction. (4) Oswestry disability index (ODI) to assess the function of back and lower limbs, (5)SF-12 for whole quality of life, (6) Pirani score to assess clubfoot deformity, and (7) foot function index to assess the impacts on quality of life due to clubfoot. Urodynamics, bladder ultrasonography, muscle strength and sensation of lower limbs will be obtained before and post treatment, to determine the patient's function of lower limbs. The investigator performing the outcome measures will be blinded to group assignment, and therefore will not participate in treatment. After randomization, the conservative group will be followed up in the outpatient clinic. The capsule surgery group will receive the nerve root axial decompression surgery.

Data Analysis: Two 2x7 MANOVAs with repeated measures will be used to examine the differences in the four measures between groups and at the five different time frames with the α level set at 0.05. Non-parametric tests (Mann-Whitney U tests) will be used to compare the differences in the urodynamics and muscle strength data over time and between groups.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged 14-20 years, without gender limitation, are willing to sign informed consent;
2. patients diagnosed with tethered cord syndrome (TCS);
3. patients accepted untethering surgery or resection of intra-lipomas or myelomeningocele after birth;
4. patients present with the recent occurrence of bladder or bowel dysfunction, with progressive deterioration, may be accompanied by motor deficits of lower extremity;
5. urodynamic examination suggests neurogenic injury;
6. the current conventional treatment is difficult to achieve satisfactory clinical outcomes.

Exclusion Criteria:

1. bladder or ureter obstruction;
2. other types of neurogenic bladder dysfunction (spinal cord injury, cerebral palsy, other brain injuries);
3. anorectal malformations;
4. poor health condition, unable to tolerate surgery;
5. patients (or their guardians) cannot give full informed consent for cognitive dysfunction;
6. patients who have participated in other clinical trials in the past 1 month.
7. patients with active hepatitis B (including HBeAg) or serological markers (HBsAg or / and HBeAg or / and HBcAb), hepatitis C, tuberculosis, cytomegalovirus infection, severe fungal infection or HIV infection;
8. patients with active peptic ulcers within 3 months before randomization.
9. patients with malignant neoplasms

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-06-16 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Changes of patient-reported scores assessing bladder function | At 1 week pre- and 1, 12, 24, 48, and 96 weeks post-operative follow-up visits.
  International Consultation on Incontinence Modular Questionnaire Short Version (ICI-Q-SF) is used to assess urinary function and the impacts on patient's quality of life due to urinary problems.

SECONDARY OUTCOMES:
Changes of patient-reported scores assessing bowel function | At 1 week pre- and 1, 12, 24, 48, and 96 weeks post-operative follow-up visits.
  Rintala Score is applied to assess bowel function and its effects on patients' quality of life.
Changes of patient-reported quality of life due to bladder dysfuction | At 1 week pre- and 1, 12, 24, 48, and 96 weeks post-operative follow-up visits.
  A new developed Chinese version of questionnaire is used to assess the quality of life in patients and parents due to bladder dysfunction.
Bladder function | At 1 week pre- and 1, 12, 48, and 96 weeks post-operative follow-up visits.
  Urodynamic testing is performed to determine the bladder function, including bladder pressure, bladder capacity, residual volume, and compliance of bladder.
Muscle power | At 1 week pre- and 1, 12, 24, 48, and 96 weeks post-operative follow-up visits.
  Muscle power is tested by manual assessment, which is classified into 6 levels.
Improvment of clubfoot deformity | At 1 week pre- and 1, 12, 24, 48, and 96 weeks post-operative follow-up visits.
  Pirani questionnaire is applied to assess the severity of clubfoot deformity by the examiner.
Changes of patient-reported scores assessing foot deformity | At 1 week pre- and 1, 12, 24, 48, and 96 weeks post-operative follow-up visits.
  Foot function index is applied to assess the impacts on patients' quality of life due to foot deformity
Changes of patient-reported scores assessing function of back and lower limbs | At 1 week pre- and 1, 12, 24, 48, and 96 weeks post-operative follow-up visits.
  Oswestry disability index (ODI) is applied to assess the function of back and lower limbs.
Changes of patient-reported quality of life | At 1 week pre- and 1, 12, 24, 48, and 96 weeks post-operative follow-up visits.
  SF-12 is applied to assess the impacts on quality of life due to tethered cord syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Jiangang Shi, MD, Study Chair — Shanghai Changzheng Hospital, Second Military Medical University
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Steinbok P, MacNeily AE, Hengel AR, Afshar K, Landgraf JM, Hader W, Pugh J. Filum Section for Urinary Incontinence in Children with Occult Tethered Cord Syndrome: A Randomized, Controlled Pilot Study. J Urol. 2016 Apr;195(4 Pt 2):1183-8. doi: 10.1016/j.juro.2015.09.082. Epub 2016 Feb 28. PMID 26926544